CLINICAL TRIAL: NCT04553783
Title: Exploration of Blood Biomarkers, Including Whole Blood Viscosity as a Prognostic Factor for Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: In Seok Lee (Other)
Responsible Party: Sponsor-Investigator, In Seok Lee, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: KC20OISI0022
Record Dates: First submitted 2020-06-03; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the usefulness of blood viscosity as a prognostic factor in patients with acute pancreatitis. The study design is a single-arm prospective cohort observational study. Blood biomarkers including blood viscosity, C-reactive protein, hematocrit, and phosphate are measured and the correlation with the severity of acute pancreatitis will be analyzed.

DETAILED DESCRIPTION:
Several scoring systems are used to evaluate the prognosis of acute pancreatitis, but they are rather complicated and clinically less useful. Blood viscosity is associated with hematocrit and inflammatory factors known to be related to the prognosis of acute pancreatitis, and our group's previous study which is not yet published showed that blood viscosity better predicts severe acute pancreatitis than other single factors such as C-reative protein. Therefore, this study aims to prospectively evaluate the usefulness of blood viscosity as a prognostic factor for acute pancreatitis. During the study period, the study is conducted on patients with acute pancreatitis between the ages of 19 and 70, and patients with acute pancreatitis after ERCP are excluded. Blood viscosities at initial and 24 hours after hospitalization, and serum phosphate, which have shown potential as a predictor of severity in post-ERCP pancreatitis in previous studies are measured. The association of these blood biomarkers with the severity of acute pancreatitis will be analyzed and compared with hematocrit, C-reactive protein, etc., which are known as a single prognostic predictor of acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-70 years old
* Acute pancreatitis

Exclusion Criteria:

* Post-Endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between 19 and 70 years of age with acute pancreatitis, excluding post-ERCP pancreatitis.
Sampling Method: Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Prediction of severity of acute pancreatitis using initial blood viscosity | 48hours after admission
  Evaluate initial blood viscosity as a predictor of the severity of acute pancreatitis

SECONDARY OUTCOMES:
Prediction of severity of acute pancreatitis using blood viscosity change after 24hours | 24hours after admission
  Prediction of severity of acute pancreatitis using blood viscosity change after 24hours
Prediction of severity of acute pancreatitis using serum phosphate | 48hours after admission
  Prediction of severity of acute pancreatitis using serum phosphate

CONTACTS AND LOCATIONS:
Overall Officials: In Seok Lee, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No